CLINICAL TRIAL: NCT00818714
Title: 0516 GCC: Stereotactic Body Radiation Therapy As A Boost After Definitive Treatment With Concurrent Chemoradiation In Patients With Non-Small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy (SBRT) as a Boost After Definitive Concurrent Chemoradiation (ChemoRT) for Non-Small Cell Lung Cancer (NSCLC) GCC 0516
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: There was no patient accrual nor study activity due to inability to fund PFTs.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040255; GCC 0516
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: IIIA, selected IIIB; (T1N2-3M0, T2N2-3M0, T3N1-3M0)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Dose escalation study to define the maximum tolerated boost dose of stereotactic body radiation therapy (SBRT) to the residual primary tumor after definitive therapy with concurrent chemotherapy and external beam radiation.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT x 3 (start 6-9 weeks following standard ChemoRT; Time between SBRT Boost treatments: 40 hours to 8 days)
  Dose Escalation Schema:
  Cohort -3: 4 Gy x3 Cohort -2: 5 Gy x3 Cohort -1: 6 Gy x3 If de-escalation is required after initial cohort
  Cohort 1: 7 Gy x 3 INITIAL COHORT Cohort 2: 8 Gy x 3 Cohort 3: 9 Gy x 3
  Continue +1 Gy x 3 until reach MTD

SUMMARY:
SBRT to deliver a boost dose to residual primary tumor after definitive doses of standard EBRT have been delivered concurrently with chemotherapy.

Serum levels of TGF-Beta1 and correlation with SBRT toxicity.

DETAILED DESCRIPTION:
This protocol is designed to use stereotactic body radiation therapy (SBRT) to deliver a boost dose to residual primary tumor after definitive doses of standard external beam radiation have been delivered concurrently with chemotherapy. It is designed to determine the toxicity profile(side effects) in the context of dose escalation of stereotactic body radiation therapy (SBRT) after definitive therapy with concurrent chemoradiation and to define the maximum tolerated dose.

Serum levels of TGF-Beta1 have been demonstrated to correlate with the incidence of the radiation toxicity, pneumonitis in patients treated with standard external beam radiation. This study will serially follow TGF-Beta1 levels in patients to see if the same correlation exists with SBRT toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of non-small cell lung cancer will be required by either biopsy or cytology. The following primary cancer types are eligible: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, bronchioloalveolar cell carcinoma, or non-small cell carcinoma not otherwise specified.
2. Eligible patients must have appropriate staging studies identifying them as specific subsets of AJCC stage III based on only one of the following combinations of TNM staging:

   * T1N2-3M0
   * T2N2-3M0
   * T3N1-3M0
   * Patients with T4 tumors (by any definition) are not eligible
3. Patients must have completed treatment with concurrent chemotherapy and external beam radiation therapy to radiation doses >59.4Gy but <70.2Gy to the primary tumor and doses >45Gy but <70.2Gy to mediastinal structures within 6 to 9 weeks of the first SBRT "Boost" treatment.
4. Patients must have had repeat staging performed after their chemoradiation and within 28 days of their first protocol treatment including: CT scan of chest and upper abdomen, FDG-18 PET scan and MRI of the brain. These studies must demonstrate no disease outside of the thorax.
5. The primary tumor must be deemed technically resectable after chemoradiation by an experienced thoracic cancer clinician, with a reasonable possibility of obtaining a gross total resection with negative margins (defined as a potentially curative resection, PCR). However, the patient must not be a candidate for PCR based on pathologic evidence of persistent mediastinal lymphadenopathy after chemoradiation or because of underlying physiological medical problems that would prohibit a PCR due to a low probability of tolerating general anesthesia, the operation, the postoperative recovery period, or the removal of adjacent functioning lung. These types of patients with severe underlying health problems are deemed "medically inoperable." Standard justification for deeming a patient medically inoperable based on pulmonary function for surgical resection of NSCLC may include any of the following: Baseline FEV1 < 40% predicted, post-operative predicted FEV1 < 30% predicted, severely reduced diffusion capacity, baseline hypoxemia and/or hypercapnia, exercise oxygen consumption < 50% predicted, severe pulmonary hypertension, diabetes mellitus with severe end organ damage, severe cerebral, cardiac, or peripheral vascular disease, or severe chronic heart disease.
6. Patients must be ≥ 18 years of age.
7. The patient's Zubrod performance status must be Zubrod 0-2.
8. Women of childbearing potential and male participants must use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills.
9. Pretreatment Evaluations Required for Eligibility include:

   * A medical history, physical examination, weight, assessment of Zubrod performance status within 2 weeks prior to study entry.
   * Evaluation by a thoracic surgeon or pulmonologist within 4 weeks prior to study entry;
   * For women of childbearing potential, a serum or urine pregnancy test must be performed within 72 hours prior to the start of protocol treatment;
   * PFTs: Routine spirometry, lung volumes, diffusion capacity, and arterial blood gases within 4 weeks prior to study entry.

   Mandatory staging studies: Must be done within 21 days prior to study entry
   * CT scan (preferably with intravenous contrast) to include the entirety of both lungs, the mediastinum, liver, and adrenal glands; Primary tumor dimension will be measured on CT.
   * Whole body positron emission tomography (PET) scan using FDG with adequate visualization of the primary tumor and draining lymph node basins in the hilar and mediastinal regions.
   * MRI of the brain
10. Patients must sign a study-specific consent form.
11. Patients must not have any serious medical or psychiatric illnesses that would prevent compliance or ability to give informed consent.
12. Labs to be within 14 days of start of SBRT:

CBC with differential, platelet count, Comprehensive metabolic panel including: electrolytes, Albumin, TBilirubin, Calcium, Cl, CO2, Creatinine, Glucose, K, TProtein, Na, BUN, AlkPhos, AST, ALT, Magnesium.

Pre-treatment laboratory values must be as follows:

WBC count: < or = 2.5 x institutional ULN; Absolute granulocyte count: > or = 1,500/mm3 Platelets: > or = 100,000/mm3 Total bilirubin: < or = 1.5 x institutional ULN Serum creatinine: < or = 1.5x institutional ULN AST and ALT: < or = 2.5 x institutional ULN Serum albumin: > or = 3.0 g/dL

Exclusion Criteria:

1 Patients with primary tumors > 5 cm or involving the central chest and structures of the mediastinum after their definitive course of chemoradiation.

2. The primary tumor of any T-stage within or touching the zone of the proximal bronchial tree defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi.

* Patients with radiographic pneumonitis obscuring clear delineation of the primary tumor or any patient who developed clinical radiation pneumonitis from their course of chemoradiation prior to protocol treatment.
* Direct evidence of regional or distant metastases after appropriate staging studies.
* Plans for the patient to receive other concomitant antineoplastic therapy (including standard fractionated radiotherapy, chemotherapy, biological therapy, vaccine therapy, and surgery). Patients may receive antineoplastic therapy at the discretion of their treating physician beginning 6 weeks after completion of protocol therapy.
* Patients with active systemic, pulmonary, or pericardial infection.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
* Major illness or psychiatric impairments, which in the investigator's opinion will prevent administration or completion of the protocol therapy and /or interfere with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity profile in the context of dose escalation of stereotactic body radiation therapy (SBRT) after definitive therapy with concurrent chemoradiation and to define the maximum tolerated dose. | Follow-up Post-SBRT: 2, 4, 6,12 weeks, every 3 months for 2 years, every 6 months for 2 years, then at the discretion of the treating M.D.

SECONDARY OUTCOMES:
To study the incidence of the radiation toxicity, pneumonitis in patients treated with SBRT by serially following TGF-Beta1 levels. | Prestudy thru post SBRT week 12

CONTACTS AND LOCATIONS:
Overall Officials: Anil Dhople, M.D., Principal Investigator — University of Maryland, Baltimore